CLINICAL TRIAL: NCT02714803
Title: Assistant Professor
Brief Title: Comparison of Different Massage Techniques Plus Conservative Applications in Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, Assistant Professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-11/33
Record Dates: First submitted 2016-03-12; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- Connective tissue massage group (Experimental): Connective tissue massage plus conservative applications including superficial thermal, electrotherapy and home exercise program were applied
  Interventions: Behavioral: "Connective tissue massage" and "Conservative applications"
- Classic massage group (Active Comparator): Classic massage plus conservative applications including superficial thermal, electrotherapy and home exercise program were applied
  Interventions: Behavioral: "Classic massage group" and "Conservative applications"
- Sham massage group (Sham Comparator): Sham massage plus conservative applications including superficial thermal, electrotherapy and home exercise program were applied
  Interventions: Behavioral: "Sham massage group" and "Conservative applications"

INTERVENTIONS:
Behavioral: "Connective tissue massage" and "Conservative applications" — Connective tissue massage and conservative aplications were applied 5 days per week for a total of 10 sessions for 2 weeks.
  Arms: Connective tissue massage group
Behavioral: "Classic massage group" and "Conservative applications" — Classic massage and conservative aplications were applied 5 days per week for a total of 10 sessions for 2 weeks.
  Arms: Classic massage group
Behavioral: "Sham massage group" and "Conservative applications" — Sham massage and conservative aplications were applied 5 days per week for a total of 10 sessions for 2 weeks.
  Arms: Sham massage group

SUMMARY:
The aim of this study is to compare of different massage techniques plus conservative aplications in low back pain treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having non specific low back pain without any relevant ongoing pathologies such as disc prolapse, spondylolisthesis, fractures, tumor, osteoporosis, infection
* Willing to participate

Exclusion Criteria:

* Spinal surgery in the past 6 months or having to undergo surgery or invasive examinations during the study;
* neurological disease;
* psychiatric disease;
* serious chronic disease that could interfere with the outcomes (e.g., cardiovascular disease, epilepsy, rheumatoid arthritis),
* pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in low back pain intensity as measured by Visual Analog Scale | Change from baseline low back pain intensity at 2 weeks

SECONDARY OUTCOMES:
Change in quality of life as assessed by Short Form-36 | Change from baseline quality of life at 2 weeks
Change in functional statue as assessed by Oswestry Disability Index | Change from baseline functional statue at 2 weeks
Change in psychologic statue as assessed by Hospital Anxiety and Depression Scale | Change from baseline psychologic statue at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk Training and Research Hospital, Ankara, Cankaya, Turkey (Türkiye)